CLINICAL TRIAL: NCT02534285
Title: the Impact of Noise on Requirements of Anesthetics During General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dresden EK30012015
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia
Keywords: Anesthesia, Inhalation; Hearing; Noise, Occupational
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Patients of the control group receive a Sham hearing protection with no effect on noise attenuation.
  Interventions: Device: hearing protection
- Intervention (Active Comparator): Patients of the Intervention group receive a Hearing protection with a noise attenuation of 20-45 decibel.
  Interventions: Device: hearing protection

INTERVENTIONS:
Device: hearing protection — Attenuation of hearing during surgery
  Other Names: PeltorTM OptimeTM III H540A, 3M, Värnamo, Sweden

SUMMARY:
The investigators hypothesize that the noise level in the operating theatre influences the patients' requirements of anesthetics. Study subject are patients undergoing abdominal surgery in combined general and epidural anesthesia. Analgesia is maintained by epidural injections of sufentanil and ropivacaine whereas general anesthesia is maintained using the inhalational anesthetic desflurane. Desflurane requirements are adjusted using neuromonitoring (BIS-Index). Intraoperative noise levels are recorded. Patients are randomized to receive hearing protections or not.

DETAILED DESCRIPTION:
All patients receive standardized anesthesia and monitoring according to the usual clinical care in the department. Placement of epidural catheters takes place before induction of general anesthesia. Thereafter, 10 ml ropivacaine 0.3% with 10 µg sufentanil are administered epidurally every 60 min to induce and maintain analgesia during surgery.

Following induction of general anesthesia and tracheal Intubation, intraoperative hypnosis is maintained using desflurane.

ELIGIBILITY:
Inclusion Criteria:

* full contractual capability
* written informed consent
* abdominal surgery in combined general/epidural anesthesia
* position during surgery: supine
* clinically normal hearing

Exclusion Criteria:

* history of psychiatric disease
* history of intraoperative awareness
* clinically impaired Hearing
* contraindication for placing an epidural catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hübler, MD, Principal Investigator — Consultant Dept. of Anesthesia; University Hospital Dresden; Technische Universität Dresden
Locations (1):
- University Hospital, Dept. of Anesthesia, Dresden, Germany

REFERENCES:
- See also: Link to the published manuscript (open access). — http://www.ai-online.info/images/ai-ausgabe/2020/06-2020/AI_06-2020_Originalia_Huebler.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from 09-04-2015 until 11-22-2016
Period: Overall Study
Arm/Group | Control | Intervention
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 22 | 39
  >=65 years | 33 | 28 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 66 (10) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 46 | 47 | 93
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Requirements of the Inhalational Anesthetic Desflurane, Measured in Expiratory Volume Percentage, to Maintain a BIS-Index Triggered Depth of Anesthesia
Description: Aimed BIS-index is 50, desflurane is measured in expiratory volume percentage
Time Frame: one hour
Measure: Mean (Standard Deviation); unit: Desflurane (Vol%)
Arm/Group | Control | Intervention
Number analyzed (Participants) | 50 | 50
Desflurane (Vol%) | 3.6 (1.2) | 3.7 (1.0)

2. Secondary Outcome: Awareness Using a Structured Interview ("Modified Brice Questionnaire")
Description: Using a structured interview ("modified Brice questionnaire") to detect episodes of intraoperative awareness
Time Frame: 1 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 months
Description: No adverse events were observed.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes